CLINICAL TRIAL: NCT03560960
Title: Multi-Center Development of a Novel Diagnostic Test for Alzheimer's Disease
Acronym: DTAD
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-37432; 1R01AG059424-01 (NIH)
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Early AD diagnosis; Pramlintide challenge test; Amyloid; Amyloid PET imaging; CSF Aβ; CSF pTau; Cognitive evaluation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Probable AD (Experimental): Participants with probable AD with positive imaging AD pathology will receive the pramlintide challenge test.
  Interventions: Drug: Pramlintide challenge test
- Amnestic MCI (Active Comparator): Participants with amnestic MCI with or without positive AD imaging pathology will receive the pramlintide challenge test.
  Interventions: Drug: Pramlintide challenge test
- Control- Normal Cognition (Active Comparator): Participants with normal cognition without any memory complaints will receive the pramlintide challenge test.
  Interventions: Drug: Pramlintide challenge test

INTERVENTIONS:
Drug: Pramlintide challenge test — Enrolled subjects will have a pre-trial blood draw (3 ml) and will be placed with an IV needle for future blood draws. Pramlintide will be subcutaneously injected in the abdominal area. For each arm the participants will be randomized so that half will be given a dose of 0.8 mcg/kg and the other half of the arm a dose of 1.6 mcg/kg. Blood will be drawn before and at 5, 30, 60, and 180 min after injection. Vital signs and blood glucose will also be checked at these time points. Thirty minutes after the injection, subjects will be offered a standard meal. Subjects will have a final check of vital signs and blood glucose approximately 15 min before discharge.
  Other Names: Symlin

SUMMARY:
In this multi-center study, the investigators plan to develop a simple blood-based test for early detection of Alzheimer's disease (AD). The test is based on a single injection of Pramlintide, an amylin analogue and FDA-approved drug currently used for treatment of diabetes. The investigative team has provided evidence in humans with full-blown AD and AD-relevant mouse models that a single injection of Pramlintide transiently renders the blood brain barrier (BBB) more permeable to Amyloidbeta (Aß) peptides, allowing their efflux from the brain compartment into the blood. This Aß efflux causes a corresponding transient elevation of blood levels of Aß, the magnitude of which the applicants believe is proportional to the brain amyloid load as determined by AV-45 PET. The measured difference in the level of plasma Aß taken just before and a short time after injection should reveal the magnitude of the transient increase in blood Aß levels.

Supportive preliminary data comes from later stage (full-blown) AD patients with more in-depth background studies in Tg2576 and 5X Familial Alzheimer's Disease (FAD) mouse models. If successful for use as an early AD biomarker (i.e., at the Mild Cognitive Impairment (MCI) stage), this could be a game-changer for both early AD diagnostics and clinical trials aimed at identifying and testing the efficacy of drugs useful for treatment of AD at early stages. If Pramlintide is effective in releasing mobile pools of Aß from the brain into the blood, this could also have some therapeutic potential, with the goal of reducing brain amyloid load.

Three groups of participants will be studied: 1) amnestic MCI with or without positive AD imaging pathology, 2) probable AD with positive imaging AD pathology, and 3) controls who have normal cognition and do not have memory complaints.

ELIGIBILITY:
Inclusion Criteria:

* Current research subjects at the BU , Memory Center VA Boston Healthcare, or Indiana University Alzheimer Disease Center
* A consensus diagnosis of probable Alzheimer's Disease (AD), amnestic mild cognitive impairment (MCI), or control
* BMI of 20-35
* Probable AD subjects must be confirmed for positive AD pathology in the central nervous center (CNS0
* Probable AD subjects must have a designated research proxy signed before they became demented.

Exclusion Criteria:

* Diabetes mellitus
* Gastroparesis
* Use of insulin, pramlintide, other injectable anti-hyperglycemic agents, such as glucagon like peptide-1 (GLP-1), or oral anti-diabetic products
* Unexplained hypoglycemia (glucose ≤ 60 mg/dL) or hyperglycemia (glucose ≥ 126 mg/dL) pre-injection
* History of stroke
* Seizures or use of anti-seizure medications
* History of brain injury and loss of consciousness
* Diagnosed cerebral amyloid angiopathy (CAA)
* Infection within 1 month

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Plasma Aβ 1-40 levels | baseline, 5, 30, 60, and 180 min after challenge test
  Plasma Aβ1-40, also known as beta-amyloid 1-40, is a biomarker measured in the blood, and it is associated with the development of Alzheimer's disease. Specifically, higher plasma concentrations of Aβ1-40, particularly when combined with lower levels of Aβ1-42, are linked to an increased risk of dementia. The normal range for Aβ 1-40 levels in human plasma is generally considered to be less than 100 pg/mL, with most studies reporting values between 30 to 60 pg/mL.
Plasma Aβ1-42 levels | baseline, 5, 30, 60, and 180 min after challenge test
  Plasma Aβ1-42, also known as beta-amyloid 1-42, is a protein fragment involved in the development of Alzheimer's disease. It is a form of amyloid-beta (Aβ) that is associated with the formation of plaques in the brain. Aβ1-42 is a key biomarker for Alzheimer's disease. Specifically, lower plasma concentrations of Aβ1-42, particularly when combined with higher levels of Aβ1-402, are linked to an increased risk of dementia. The reference interval for plasma Aβ1-42 levels in cognitively normal subjects is typically between 8.12 and 29.00 pg/mL.
Plasma Aβ and t-tau changes | baseline, 5, 30, 60, and 180 min after challenge test
  Plasma total tau (t-tau) levels can indicate subclinical brain and cognitive deficits, potentially predicting the risk of neurodegenerative conditions in normal aging. Higher plasma t-tau levels have been associated with poorer cognitive function, reduced glucose uptake, thinning of the temporal lobe, and even increased risk of all-cause dementia. The reference range for plasma total tau (t-tau) is typically reported as 0.20-3.12 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Qiu, MD PhD, Principal Investigator — Boston Medical Center and BUSM
Locations (3):
- United States (3):
  - Indiana University Alzheimer Disease Center, Indianapolis, Indiana
  - BU Alzheimer Disease Center, Boston, Massachusetts
  - Memory Center VA Boston Healthcare, Jamaica Plain, Massachusetts

IPD SHARING:
Plan to Share IPD: No